CLINICAL TRIAL: NCT04121962
Title: Pilot Peer Mentor Intervention to Train Black MSM to Use and Promote Home-based HIV and STI Testing
Brief Title: A Pilot Peer Mentor Intervention That Trains Black Men Who Have Sex With Men (BMSM) to Use and Promote Uptake of HIV/STI Self-Testing to Peers and Sex Partners: STAR Study (Self-Testing at Your Residence)
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R34MH118178 (NIH); IRB00009216 (Other: JHSPH IRB)
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: HIV/AIDS; Sexually Transmitted Diseases
Keywords: Black MSM; Social network
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Mentor (Experimental): Peer Mentor Training is 5 individual sessions with a 30 day check-in session. This condition is focused on training Index with communication skills to promote HIV and STI testing and treatment and pre-exposure prophalaxis (PrEP) to individuals in their social networks. Peer Mentor training is conducted by a one health educator. The sessions are held once a week and will last approximately 60 minutes.
  Interventions: Behavioral: Peer Mentor
- Control (Active Comparator): Is one individual-based session which will be conducted by sending a video about the website of a health educator.
  Interventions: Behavioral: Website only

INTERVENTIONS:
Behavioral: Peer Mentor — Participants will be trained to be Peer Mentors and promote home-based testing to their social network
  Arms: Peer Mentor
Behavioral: Website only — Participants will be given instructions on how to use the project website to request kits to test for HIV at home and collect specimens for lab testing.
  Arms: Control

SUMMARY:
The objectives of the study are to assess the feasibility, reach and preliminary efficacy of a brief intervention that trains Black men who have sex with men [referred to as Index] (a) to use home-based testing for HIV and sexually transmitted infections and (b) promote home-based testing to their peers and sexual partners.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) increase one's risk of HIV infection, are serious co-infections that affect HIV clinical outcomes, and remain a risk for individuals using PrEP. Self-testing methods address barriers to clinic-based testing by offering convenience and privacy and have been shown to be well accepted by MSM. Therefore, use of self-testing is a potential approach through which to improve HIV and STI testing rates in MSM. Internet-based distribution (herein: web-based) of STI self-test kits enables an individual to request sampling kits via a website, mail biological specimens (e.g. urethral swabs) to a laboratory for testing, and view test results through a web-based account. Web-based self-HIV oral testing enables an individual to request a test kit, collect an oral specimen, and receive results within 20 minutes. Despite these potential benefits and reports of willingness to use free self-testing, uptake has been low due to barriers such as concerns about accuracy of the tests, apprehension to collect specimens, low risk perception, and the desire for counseling. In the proposed study, investigators will pilot test an intervention that address these barriers by training BMSM with information about the accuracy of the HIV rapid oral test kit, demonstrating how to properly collect specimens for HIV and STIs (gonorrhea, chlamydia and syphilis) self-testing, and providing resources for linkage to HIV and STI treatment and PrEP services. Study participants will utilize a secure website to request test kits.

ELIGIBILITY:
Inclusion Criteria:

* self-report male sex
* condomless anal sex with >1 male in the prior 6 months
* self-report Black race
* aged 18 or older
* internet use at least once a week.

Exclusion Criteria:

* younger than 17

Ages: 17 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Biologic male who identifies as male
Enrollment: 163 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin E Tobin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighthouse Studies @ Peer Point, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share data in a way that will protect participant confidentiality. Within 12 months of publication of the primary papers for this study, a dataset of aggregate values will be made available. Due to the highly sensitive nature of the data collected and the characteristics of this often stigmatized population, no client-level data will be shared until the entire cohort is accrued and completed, even that which is de-identified; this will reduce the risk of small numbers resulting in deductive identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after data collection is over
Access Criteria: To Be Determined

REFERENCES:
- [Background] Tobin KE, Heidari O, Winiker A, Pollock S, Rothwell MD, Alexander K, Owczarzak J, Latkin C. Peer Approaches to Improve HIV Care Cascade Outcomes: a Scoping Review Focused on Peer Behavioral Mechanisms. Curr HIV/AIDS Rep. 2022 Aug;19(4):251-264. doi: 10.1007/s11904-022-00611-3. Epub 2022 Jul 7. PMID 35798989

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 163 participants were consented. 64 participants assigned to Peer Mentor condition (Index and network); 55 participants assigned to the control (Index and network); 44 participants were withdrawn pre-assignment and not assigned to a condition.
Groups:
- Peer Mentor: Peer Mentor Training is 5 individual sessions with a 30 day check-in session. This condition is focused on training Index with communication skills to promote HIV and Sexually Transmitted Infection (STI) testing and treatment and pre-exposure prophalaxis (PrEP) to individuals in their social networks.
  Peer Mentor training is conducted by a one health educator. The sessions are held once a week and will last approximately 60 minutes.
- Control: Participants will receive information on how to use the website to request at-home test kits
  Website only: Participants will be given instructions on how to use the project website to request kits to test for HIV at home and collect specimens for lab testing.
Period: Overall Study
Arm/Group | Peer Mentor | Control
Started | 64 | 55
Completed | 22 | 16
Not Completed | 42 | 39
Not completed — Lost to Follow-up | 42 | 39

BASELINE CHARACTERISTICS:
Population: Participants who were consented
Groups:
- Not Assigned: Participants not randomized to either condition
- Total: Total of all reporting groups
Arm/Group | Peer Mentor | Control | Not Assigned | Total
Number analyzed (Participants) | 64 | 55 | 44 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 55 | 44 | 163
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 38.0 (10.6) | 38.5 (9.20) | 35.25 (3.70) | 38.2 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 62 | 54 | 44 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 2 | 10
  Not Hispanic or Latino | 59 | 52 | 42 | 153
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 57 | 53 | 2 | 112
  White | 1 | 1 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 41 | 44

OUTCOME MEASURES:

1. Primary Outcome: Session Attendance
Description: number of participants who completed 80%
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentor | Control
Number analyzed (Participants) | 64 | 55
Participants | 64 | 55

2. Primary Outcome: Number of Index Participants Who Requested Test Kits
Description: Number of Index participants who requested test kits is reported
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentor | Control
Number analyzed (Participants) | 64 | 55
Participants | 9 | 17

3. Primary Outcome: Number of Participants Who Return Kits for Testing
Description: Number of participants who returned kits to lab for testing is reported.
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentor | Control
Number analyzed (Participants) | 64 | 55
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants who were not assigned to a condition were not assessed for adverse events.
Arm/Group | Peer Mentor | Control
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/55
Other Adverse Events (participants affected / at risk) | 0/64 | 0/55

LIMITATIONS AND CAVEATS:
This study occurred during the COVID-19 pandemic and amid the stay at home orders. Therefore recruitment was interrupted and the delivery of the intervention and control were remote. The stay-at home orders also disrupted the follow-up activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04121962/Prot_SAP_000.pdf